CLINICAL TRIAL: NCT06701331
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety and Efficacy of Upadacitinib in Combination With Topical Corticosteroids in Children From 2 to Less Than 12 Years of Age in Japan With Moderate to Severe Atopic Dermatitis
Brief Title: Safety and Efficacy of Upadacitinib in Combination With Topical Corticosteroids in Children From 2 to Less Than 12 Years of Age in Japan With Moderate to Severe Atopic Dermatitis
Acronym: Start Up Japan
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M25-145
Record Dates: First submitted 2024-11-21; First posted 2024-11-22 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
Keywords: Upadacitinib
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo / Upadacitinib + Topical Corticosteroids (TCS) (Placebo Comparator): Participants will receive placebo orally once a day (QD) in combination with TCS for 12 weeks in the double-blind treatment period. At Week 12 participants will then be switched to receive open-label upadacitinib daily adult equivalent dose in combination with TCS.
  Interventions: Drug: Placebo; Drug: Upadacitinib
- Upadacitinib + Topical Corticosteroids (TCS) (Experimental): Participants will be randomized to receive the upadacitinib daily adult equivalent dose in combination with TCS once a day (QD) during the double-blind and open label treatment periods for a total of 52 weeks
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo — Tablets taken orally once a day (Or equivalent oral solution taken two times a day)
  Other Names: ABT-494; RINVOQ®
  Arms: Placebo / Upadacitinib + Topical Corticosteroids (TCS)
Drug: Upadacitinib — Tablets taken orally once a day (Or equivalent oral solution taken two times a day)
  Other Names: ABT-494; RINVOQ®

SUMMARY:
Pediatric atopic dermatitis (AD), also known as childhood eczema, is a skin condition that may cause a rash and itching due to inflammation of the skin. The purpose of this study is to assess the change in disease activity (Efficacy) and to assess the safety of upadacitinib in combination with topical corticosteroids (TCS) in pediatric participants 2 to 11 years of age in Japan with moderate to severe AD who are candidates for systemic therapy.

Upadacitinib is approved for the treatment of moderate to severe AD in adults and adolescents 12 years of age and older in many countries, including Japan. This study comprises a 35-day screening period; a 12-week, randomized, double-blind treatment period where there will be a 1 in 2 chance that a participant is assigned placebo. This will be followed by an open-label upadacitinib treatment period up to Week 52.

Around 98 participants will be enrolled in the study at approximately 35 sites in Japan.

Participants will receive upadacitinib oral tablets, or matching placebo, once daily (or an adult equivalent oral solution dose twice a day) for up to 52 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care . Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by clinical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* A minimum weight of 10 kg and weight and height ≥ -2.0 SD for their age according to Japanese standard growth charts at the Baseline visit.
* Atopic Dermatitis (AD), according to Hanifin and Rajka criteria, with onset of symptoms at least 6 months prior to Baseline.
* Eczema Area and Severity Index (EASI) score ≥ 16; validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) score ≥ 3; ≥ 10% body surface area (BSA) of AD involvement at the Baseline visit; and Baseline weekly average of daily WIS or WSI-NRS ≥ 4.
* Participant has applied a topical, additive-free, bland emollient or moisturizer twice daily for at least 7 days before the Baseline visit.
* Documented history (within 6 months of the Baseline visit) of inadequate response or intolerance to topical corticosteroids (TCS) and/or topical calcineurin inhibitors (TCI) or a systemic immunomodulating therapy, or medical inadvisability of available systemic therapy (e.g., because of important side effects or safety risks).

Exclusion Criteria:

* Participants that have current and/or history of other active skin diseases (e.g., psoriasis or Netherton syndrome or lupus erythematosus) or skin infections (bacterial, fungal, or viral) requiring systemic treatment within 4 weeks of the Baseline visit or that would interfere with the appropriate assessment of AD lesions.
* Participants that have used topical treatments for AD (except for topical emollient or moisturizer treatments) including but not limited to TCS, TCI, or topical PDE-4 inhibitors, within 7 days of the Baseline visit or any the following prohibited AD treatments within the specified timeframes below prior to the Baseline visit:

  * Systemic therapy for AD, including but not limited to corticosteroids and cyclosporine, within 4 weeks;
  * Targeted biologic treatments within 5 half-lives (if known) or within 12 weeks, whichever is longer;
  * Phototherapy treatment, laser therapy, tanning booth use, or extended sun exposure that could affect disease severity or interfere with disease assessments within 4 weeks.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Estimated)
Dates: Start 2024-12-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Eczema Area and Severity Index (EASI) 75 | At Week 12
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1],
  An EASI 75 response is defined as a 75% reduction (improvement) from Baseline in EASI score.
Number of Participants With Adverse Events | From first dose of study drug until 30 days following last dose of study drug (up to approximately 56 weeks)
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not the event is considered causally related to the use of the product.

SECONDARY OUTCOMES:
Percentage of participants achieving validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) 0/1 with a reduction from Baseline of ≥ 2 points | At Week 12
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
Percentage of participants achieving an improved (reduced) weekly average Worst Itch Scale (WIS) score of ≥ 4 from Baseline for participants equal or greater than 6 years old with a weekly average WIS of ≥ 4 at Baseline | At Week 12
  The WIS is an assessment tool that participants use to report the intensity of their pruritus. Using an 11-point scale (0 to 10) where 0 indicates no itching and 10 indicates worst itching possible, participants are asked 2 questions: "What was the worst itch you had today?" and "What was the worst itch you had last night?" The WIS will be administered to participants ≥ 6 years of age at the time of the Baseline visit.
Percentage of participants achieving an improved (reduced) weekly average Worst Scratch/Itch numerical rating scale (WIS-NRS) score of ≥ 4 from Baseline for participants less than 6 years old with a weekly average WIS of ≥ 4 at Baseline | At Week 12
  The WSI-NRS is an assessment tool that evaluates a participants scratching and itching intensity at its worst in the past 24 hours as assessed by the participants parent/legally authorized representative. Intensity is assessed on an 11-point scale (0 to 10) where 0 indicates no scratching/itching and 10 indicates worst scratching/itching possible.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (25):
- Japan (25):
  - Central Clinic /ID# 269205, Nagoya, Aichi-ken
  - Fujita Health University Hospital /ID# 269201, Toyoake, Aichi-ken
  - Miyata Dermatology Clinic /ID# 269200, Matsudo-Shi, Chiba
  - Hoshikuma Dermatology ・ Allergy Clinic /ID# 270192, Fukuoka, Fukuoka
  - Saruta Dermatology Clinic /ID# 270416, Fukuoka, Fukuoka
  - Tokunaga Skin Clinic /ID# 270189, Kasuga-shi, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Japan /ID# 269206, Kitakyushu-shi, Fukuoka
  - Gunma University Hospital /ID# 272319, Maebashi, Gunma
  - Sapporo Shiroishi Dermatology Clinic /ID# 269691, Sapporo, Hokkaido
  - Hirase Allergie Children's Clinic /ID# 271208, Kobe, Hyōgo
  - Ryuseidai Children's Clinic /ID# 271400, Tsukuba, Ibaraki
  - University of Tsukuba Hospital /ID# 271238, Tsukuba, Ibaraki
  - Takeoka Dermatology Clinic /ID# 269199, Marugame, Kagawa-ken
  - Musashikosugi Sasamoto Pediatric and Allergy Clinic /ID# 270381, Kawasaki-shi, Kanagawa
  - National Hospital Organization Sagamihara National Hospital /ID# 271575, Sagamihara, Kanagawa
  - Aoi Dermatology Clinic /ID# 274265, Kamimashiki-gun, Kumamoto
  - Medical corporation Kojinkai Yoshioka Dermatology Clinic /ID# 269198, Neyagawa, Osaka
  - Hayami Dermatology Clinic /ID# 269945, Osaka, Osaka
  - Momodani Skin Clinic /ID# 270384, Osaka, Osaka
  - Medical corporation Jun Dermatology Clinic /ID# 269953, Osaka, Osaka
  - Dermatology and Ophthalmology Kume Clinic /ID# 271854, Sakai, Osaka
  - Dokkyo Medical University Hospital /ID# 270367, Mibu, Tochigi
  - Fukuwa clinic /ID# 269203, Chuo-ku, Tokyo
  - Seijo Sasamoto Pediatric Allergy Clinic /ID# 270194, Setagaya-ku, Tokyo
  - Saitama City Hospital /ID# 271392, Saitama

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-145